CLINICAL TRIAL: NCT03387618
Title: Feasibility Assessment of Next-generation PET Technology and Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Ohio Third Frontier (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017H0119/RP0506
Record Dates: First submitted 2017-11-20; First posted 2018-01-02 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: New-generation Digital PET/CT Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Investigational Scan (Experimental): new-generation digital PET/CT imaging technology
  Interventions: Diagnostic Test: Digital PET/CT imaging

INTERVENTIONS:
Diagnostic Test: Digital PET/CT imaging — Next generation PET/CT imaging

SUMMARY:
The purpose of this study is to assess the feasibility of investigational Positron Emission Tomography (PET) imaging using the new generation digital detector PET technology for new procedures beyond the current standard of care.

DETAILED DESCRIPTION:
The objectives of this study are:

1. To enable innovative PET imaging in association with a clinical trial to add potential future biomarker readouts for disease characterization and therapy management.
2. To generate preliminary and comparative imaging data for potential confirmatory clinical trials using innovative imaging timepoints, acquisition, dose, and timing approaches, and/or postprocessing procedures.
3. To explore digital PET imaging for new indications where PET is not currently considered a standard of care diagnostic procedure in order to be able to design future clinical trials.

PET imaging is increasingly being used as a diagnostic modality in cancer detection and staging, neuro-molecular assessment, cardiovascular-molecular imaging, physiological/musculoskeletal imaging, and response assessment. Additionally, PET imaging is utilized in the detection and assessment of inflammatory processes. Constant advances in detector technology, image acquisition, and post-processing approaches could lead to the increased utility of PET in many currently unmet clinical scenarios.

The investigators have already performed an intra-individual comparison trial demonstrating advanced capabilities of digital PET technology in regard to lesion detection, lesion characterization, quantification, duration of scan time, and reduction of radiation dose. The digital PET is now fully FDA approved, and in this trial the investigators need to generate preliminary data in order to design prospective clinical trials that allow the validation of a hypothesis. The investigators have demonstrated the safety of the system [now FDA approved] and the overall efficacy in relation to current clinical care practice standards; however, the technology enables the change of those standards for which the investigators need to demonstrate the clinical feasibility that they have either shown in pre-clinical PET imaging or via simulations.

This research focuses on evaluating the new capabilities of PET imaging which may be improved or enabled by a new generation of fully digital PET systems. In order to change clinical practice, the investigators need to first generate data on the potential capabilities of this major technology improvement. The investigators will be performing and evaluating investigational PET/CT imaging beyond the current standard of care practice. Prior studies by the study team have already performed comparisons between the new and current PET imaging; however, the digital PET studies were constrained by being performed as a comparison to standard of care. In this clinical trial, the investigators can conduct research studies at innovative time points or using innovative procedures currently not covered by insurance, such as repeat imaging prior to treatment or midway through treatment for replanning purposes or to find better quantitative readouts to improve diagnosis and disease management. The investigators intend to conduct PET imaging also for indications not typically covered by insurance, such as cardiac, neuro-related, or orthopedic/sports medicine indications. The investigators may also perform imaging with FDA approved radiotracers beyond their normal use (off-label) to explore the synergistic capabilities of the new generation of PET imaging.

This prospective study will utilize investigational PET acquisitions on the newly available digital photon counting detector platform to develop and optimize PET acquisition and postprocessing techniques as well as to generate preliminary and comparative data for potential confirmatory clinical trials. The investigators will assess these innovations in regard but not limited to visual inspection of lesions, normal tissue, sentinel nodes and imaging artifacts, semi-quantitative and blinded reader analysis. The PET methodologies that are planned to be used as part of this study will allow the investigators to obtain morphological, functional and molecular information in ways beyond any current standard of care imaging procedures.

Patients are anticipated to be recruited from 3 general populations. 1 - Patients enrolled in a clinical trial where innovative PET imaging may be beneficial to the trial, although not necessarily the individual patient. This would include patients enrolled in a clinical trial exploring a new treatment approach for whom imaging at other timepoints in treatment would not be covered by insurance and therefore not considered standard of care (SOC). 2 - Any patient with a concern for a medical condition / question not yet fully resolved by SOC practice for whom a treating physician believes that a research PET may have a potential to address the medical question and help for future patients with similar questions. For example, this could include a patient presenting with heel pain for whom standard x-ray shows no confirmation of injury, but the physician feels an innovative PET bone scan could help identify the cause of the pain. 3 - Any patient having a SOC PET scan who would be interested in receiving an investigational scan, either as part of or in addition to the SOC scan. This would include patients already scheduled for a SOC scan who would be willing to have an investigational PET acquisition immediately following the standard acquisition for example acquired with a shorter scan time. This would also include patients who have already had a SOC PET examination, but would be willing to have a second, investigational PET exam, with a significantly reduced radiotracer dose for example.Thus the radiation dose and exposure associated with the investigational imaging would be in addition to any standard of care imaging, although the two will be combined whenever appropriate.

Patients will be asked to provide study personnel with authorization to access their medical records for follow-up on future related procedures as well as the current outcome of their standard of care imaging. Additionally, participants will be asked if their imaging data from this study can be used in a de-identified manner in the future for comparison with other imaging data or as preliminary data for the protocol development of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers greater than or equal to 18 years of age having a medical diagnosis which justifies exploratory PET imaging

Exclusion Criteria:

* Participants who are pregnant or lactating
* Prisoners
* Subjects incapable of giving informed written consent or who are unlikely to complete the imaging procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2017-09-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Image Quality | through study completion, an average of 3 years
  Assessing the benefit of the new advanced PET technology to improve the capabilities of PET imaging
Accelerated Acquisition Time | through study completion, an average of 3 years
  The necessary time of the patient to be on the imaging system table/bed will be measured and reported. Currently, the common acquisition time is approximately 20 minutes. We explore to reduce imaging times to 5 or 10 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Martha Morehouse Medical Plaza, Columbus, Ohio, United States

DOCUMENTS (2):
  • Study Protocol (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT03387618/Prot_000.pdf
  • Informed Consent Form (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT03387618/ICF_001.pdf